CLINICAL TRIAL: NCT04591288
Title: Functional Electrical Stimulation (FES) to Improve Gait in CP Short Title
Brief Title: FES to Improve Gait in CP
Acronym: CP FES Walking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by the sponsor for not fully meeting subject recruitment targets.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Samuel C.K. Lee, PhD, PT, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PHL1809
Record Dates: First submitted 2019-08-20; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Palsy; Spastic Diplegia Cerebral Palsy; Gait
Keywords: Cerebral Palsy; Functional electrical stimulation; Neurotherapeutic
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled two-treatment group clinical trial. We randomly assign subjects to either an FES-Treadmill group, a Treadmill-Only group, or a Control group. The FES-Treadmill group will undergo an FES-assisted treadmill training protocol. The Treadmill-Only group will undergo the same protocol without FES assistance. The control group will not receive treatment. Additionally, following their "no-treatment" period, we will randomize control group subjects into one of the two treatment groups. This design allows us greater power to identify treatment group differences while accommodating parents who might ordinarily not want their child to participate in a non-treatment group. Initially, each group will consist of 14 subjects. Following crossover, the FES-Treadmill and Treadmill-Only groups will consist of 21 subjects while the control group remains 14 subjects.
Who Masked: Outcomes Assessor
Masking Description: All the clinical assessments will be performed by masked Physical Therapist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FES + Treadmill (Experimental): Functional Electrical stimulation walking group.
  Interventions: Other: Functional Electrical Stimulation protocol
- Treadmill only (Active Comparator): Treadmill walking group (no electrical stimulation).
  Interventions: Other: Treadmill only protocol
- Control (No Intervention): Control group.
  After control period of 12 weeks, they are randomized into FES + Treadmill or Treadmill group.

INTERVENTIONS:
Other: Functional Electrical Stimulation protocol — FES-assisted treadmill walking followed by a 12-week follow-up period. Subjects will train three times a week walking at a target speed corresponding to 60-80% of their age-predicted maximum heart rate. Each training session will consist of five six-minute walking bouts, with five-minute rest periods between bouts. Each treadmill bout consists of alternating one- minute intervals of FES on and FES off. For the last walking bout, the first three minutes will be FES-assisted on the treadmill and the last three minutes will be overground walking without FES assistance to promote carryover effects. Total walking time is 30 minutes and the entire training session lasts approximately 50 minutes.
  Arms: FES + Treadmill
Other: Treadmill only protocol — We will implement a 12-wk Treadmill training protocol consisting of treadmill walking followed by a 12-week follow-up period. Subjects will train three times a week walking at a target speed corresponding to 60-80% of their age. Each training session will consist of five six-minute walking bouts, with five-minute rest periods between bouts. Total walking time is 30 minutes and the entire training session lasts approximately 50 minutes.
  Arms: Treadmill only

SUMMARY:
The goal of this proposal is to mitigate the typical decline in walking function experienced by children with cerebral palsy (CP) via a Functional Electrical Stimulation (FES)-assisted treadmill training intervention.

In this study, the investigators intend to use thier CP FES Gait Training System to assess the neurotherapeutic effects of an FES-assisted treadmill training intervention on walking performance in children with CP. The research design consists of a randomized, controlled, two-treatment study in which the control subjects will cross-over into one of the two treatment groups. An FES-assisted training group will undergo twelve weeks of FES-assisted treadmill training using a distributive practice protocol consisting of alternating bouts of walking with and without FES assistance, followed by over ground walking reinforcement. A treadmill-only training group will undergo the same training regimen without FES-assistance. Finally, a non-intervention group will serve as a control. The investigators will analyze treatment efficacy via functional and biomechanical and measures collected pre-training, post-training and after a twelve-week follow-up period.

DETAILED DESCRIPTION:
Aim 1: Assess the neurotherapeutic effects of FES-assisted treadmill and treadmill-only training on walking function relative to each other and to the control group.

1.1 The FES-assisted treadmill and treadmill-only groups will demonstrate greater improvements in walking speed and walking distance than the control group post-training and at follow-up. The FES-assisted treadmill group will show greater improvements than the treadmill-only group.

1.2 The FES-assisted treadmill and treadmill-only groups will demonstrate greater improvement in walking energy efficiency than the control group post-training and at follow-up. The FES-assisted treadmill group will show greater improvement than the treadmill-only group.

1.3 The FES-assisted treadmill and treadmill-only groups will demonstrate greater improvements in GMFM, perceived functional mobility, quality of life and self-perception measures than the control group post-training and at follow-up. The FES-assisted treadmill group will show greater improvements than the treadmill-only group.

Aim 2: Assess the differential neurotherapeutic effects of FES-assisted treadmill and treadmill-only training on walking biomechanics. The investigators will measure these effects using instrumented motion capture.

2.1 The FES-assisted treadmill group will demonstrate greater improvements in gait kinematics in stance phase (higher peak hip and knee extension and lower peak ankle dorsiflexion) and swing phase (higher peak knee extension and larger knee excursion) than the treadmill only and non-intervention groups 2.2 The FES-assisted treadmill group will demonstrate greater improvements in lower extremity kinetics (lower hip and knee extensor moments and increased ankle plantarflexion power) than the treadmill only and non- intervention groups.

2.3 The FES-assisted treadmill group will demonstrate greater improvements in spatiotemporal gait parameters (increased step length and gait velocity, decreased step width and double support time) than the treadmill- only and control groups.

Aim 3: Identify predictive measures of training efficacy. 3.1 Pre-training walking speed and energy efficiency will correlate with improvements in walking performance measures of Aim 1.

3.2 Increased neuroprosthetic correction of gait biomechanics measures achieved by FES will be positively correlated with walking performance measures of Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18
* Diagnosis of spastic diplegic CP
* Gross Motor Functional Classification Scale (GMFCS) level I-III
* Hip migration < 40%
* Displays crouch, equinus, or jump type gait
* At least 0° passive dorsiflexion range of motion (can come to a neutral position)
* Sufficient visuoperceptual, cognitive and communication skills
* Seizure-free or well-controlled seizures
* No other neurological or musculoskeletal disorders (e.g. dystonia, severe scoliosis, hip instability)
* Ability to travel to University of Delaware or Shriners Hospital for children multiple times per week for training and assessment
* Ability to communicate pain or discomfort
* Ability to consent (if 18 years old) or obtain parent/guardian consent (if under 18)

Exclusion Criteria:

* Diagnosis of athetoid or ataxic CP
* Scoliosis with primary curve > 49%
* Spinal fusions extending into pelvis
* Lower Extremity (LE) joint instability or dislocation
* Severe tactile hypersensitivity
* LE botulinum (Botox) injections in the past 6 mo.
* Implanted medical device contraindicative of FES
* Pregnancy
* Severe LE spasticity (Modified Ashworth Scale score of 4 or greater)
* History of pulmonary disease limiting exercise tolerance (Asthma Control screen)
* History of cardiac disease (AHA screen)
* Excessive LE joint pain during walking
* Severely limited joint range of motion / irreversible muscle contractures, i.e.> 10°knee flexion, >15° hip flexion contractures, or >5° plantarflexion contractures
* LE surgery or significant injury within 1 yr.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle Tone | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  We use the Modified Ashworth Scale to measure resistance to passive movement about a joint with varying degree of velocity (Muscle tone/spasticity). Score ranges from 0-4, with 6 choices where score of 0 means no increase in tone and score of 4 means rigid limb with no flexion or extension. Our training approach using repetitive electrical stimulation may also lower spasticity, which can also facilitate improved functional mobility.
Walking Speed | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Walking speed is an indicator of functional mobility. By our training methods, we hypothesize making improvements in motor learning and gait biomechanics. Improved walking speed would indicate that such improvements have occurred.
Walking Distance | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Walking distance (in a fixed period of time) is an indicator of endurance. Improved motor learning and gait biomechanics from our training methods would improve gait efficiency and thus, endurance.
Energy Expenditure | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Energy expenditure is a measure of cardiovascular fitness and walking efficiency.
  By means of exercise at 60-80% max heart rates, it is expected that cardiovascular fitness would improve. Energy expenditure measurements allow for measurement of cardiovascular fitness.
Gross Motor Function Measure | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Gross Motor Function Measure (GMFM) is a measure of motor function that indicates disablement. Improved motor control and gait biomechanics from training should be reflected in overall gross motor function, which is assessed via the GMFM.
Balance Evaluation Systems Test | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Balance Evaluation Systems Test (BESTest) is a measure of balance function. The BESTest will allow for assessing the impact of anticipated improvements in motor control and gait biomechanics from training on balance.
Timed Up-And-Go | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Timed Up-And-Go (TUG) is a measure of functional mobility and will allow for assessing the impact of anticipated improvements in motor control and gait biomechanics.
Instrumented Gait Analysis | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Joint Kinematics
Electromyography | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Muscle activation timing measured with electromyography during gait analysis allows for mechanistic study of anticipated improvements in motor control and gait as well as comparison to typical norms.
Activities-Specific Balance Scale | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  The Activities-Specific Balance Scale (ABC Scale) survey allows measurement of perceived functional mobility by assessing balance confidence to perform daily activities of living without falling. 16 items are rated on a rating scale with range of 0-100. Score of 0 means no confidence and 100 means complete confidence. Average score of 16 items is the overall score. Such measures will assess the impact of anticipated improvements in motor control and gait bio-mechanics from training.
Participation in Life Events | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Participation in life events (LIFE-H) survey measures how much a person is engaging or participating with their peers and community. Weighted score ranges between 0-10 with 0 score being no accomplishment and 10 means complete accomplishment. Such measures will assess the impact of anticipated improvements in motor control and gait biomechanics from training.
Self-Perception | Three assessment points in time: a Pre Assessment before beginning training (Week 1), a Post Assessment following training (Week 14), and a Follow-Up Assessment twelve weeks after completion of training (Week 27).
  Self-Perception (Piers-Harris-2) survey measures physical and emotional well-being and self-esteem and will allow assessment of the impact of anticipated improvements in motor control and gait biomechanics from training.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel CK Lee, Ph.D., Principal Investigator — University of Delaware
Locations (2):
- United States (2):
  - University of Delaware, Newark, Delaware
  - Shriner's Hospital for Children, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The proposed experiments will generate data for publications in high quality peer reviewed journals. We will also present our findings at national meetings of neurorehabilitation scientists and clinicians and neuroscience and motor control meetings. To have the most impact, it is important that we present our findings to both clinicians and scientists, therefore, in addition to these standard approaches, we will seek out regular opportunities to present both the rationale and results of our work to local and regional clinicians as well as local and regional stroke support groups.
  Once the primary hypotheses of the current proposal are tested, all data will be de-identified and be deposited in the DASH (The Data and Specimen Hub) repository.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol and data will be shared on publication of primary results

REFERENCES:
- See also: Principal Investigator's Webpage — https://sites.udel.edu/pt/dr-samuel-lee/